CLINICAL TRIAL: NCT05286320
Title: Phase Ib/II Trial of Combining Pembrolizumab and Lenvatinib With Stereotactic Body Radiotherapy for Hepatocellular Carcinoma Patients With Portal Vein Thrombosis.
Brief Title: Phase Ib/II Trial of Combining Pembrolizumab and Lenvatinib With SBRT for HCC Patients With Portal Vein Thrombosis.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202108042MIPA
Record Dates: First submitted 2022-02-06; First posted 2022-03-18 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2022-09

CONDITIONS: Unresectable Hepatocellular Carcinoma; Pembrolizumab; Lenvatinib; Stereotactic Body Radiotherapy
Keywords: Unresectable Hepatocellular Carcinoma; Immunotherapy; Stereotactic body radiotherapy; targeted therapy
MeSH Terms: interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Target-/Immuno-therapy for advanced HCC w PVTT Lenvatinib/Pembrolizumab plus SBRT combinations (Experimental): Five-fraction SBRT (week 4-week 5) to PVTT and connected HCC tumor in 2 weeks Lenvatinib 12/8 mg/day for 96 weeks (no lenvatinib from 7 day before SBRT to 7 days after SBRT) Pembrolizumab 200 mg q 3 week x 32 cycles
  Interventions: Drug: Lenvatinib/Pembrolizumab plus SBRT combinations

INTERVENTIONS:
Drug: Lenvatinib/Pembrolizumab plus SBRT combinations — Five-fraction SBRT (week 4-week 5) to PVTT and connected HCC tumor in 2 weeks Lenvatinib 12/8 mg/day for 96 weeks (no lenvatinib from 7 day before SBRT to 7 days after SBRT) Pembrolizumab 200 mg q 3 week x 32 cycles
  Other Names: Lenvima; Keytruda

SUMMARY:
HCC patients with PVTT (main trunk or the first-degree branch) treated with the combination of pembrolizumab (Ketruda), lenvatinib (Lenvima), and SBRT.

DETAILED DESCRIPTION:
Protocol treatment includes : Pembrolizumab is intravenously infused every 3 weeks and lenvatinib is orally given every day for a total of 2 years. SBRT (5 fractions within 17 days) to the PVTT and adjacent connecting HCC tumor is delivered in the second cycle of pembrolizumab, with the discontinuation of lenvatinib 7 days before and after SBRT.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 20 years of age on the day of signing informed consent with histologically confirmed diagnosis of HCC or those diagnosed by the EASL non-invasive criteria for HCC will be enrolled in this study.
2. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 220 days after the last dose of study treatment and refrain from donating sperm during this period.
3. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 150 days after the last dose of study treatment.
4. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
5. Have measurable disease based on mRECIST.
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
7. Have adequate organ function as defined in the following criteria (Specimens must be collected within 10 days prior to the start of study intervention) :(1)Absolute neutrophil count (ANC) ≥1500/µL. (2)Platelets ≥100000/µL. (3)Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L. (4)Creatinine OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN. (5)Total bilirubin ≤1.5 ×ULN (mg/dL) OR direct bilirubin ≤ULN for participants with total bilirubin levels >2.5 × ULN (mg/dL).(6)AST (SGOT) and ALT (SGPT) ≤5 × ULN. (7)Alkaline phosphatase ≤2 × ULN.(8)Child-Pugh class Class A. (9)International normalized ratio (INR) OR prothrombin time (PT)、Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
8. Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening. Participants must have completed curative anti-viral therapy at least 4 weeks prior to starting study intervention. Participants with HBV will be eligible as long as they meet the following criteria: (1) Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to starting study intervention. (2)Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
9. Patients have PVTT in the main trunk (VP4) or central branch (VP3).
10. Previous liver resection, embolization, or ablative therapy is permitted.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to [allocation]. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-HCC therapy including investigational agents or other local therapy within 4 weeks prior to [allocation].
4. Has received prior radiotherapy to non-liver sites within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive or modulation therapy within 7 days prior to the first dose of study drug.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
8. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
9. Has severe hypersensitivity (≥Grade 3) to pembrolizumab/Lenvatinib and/or any of their excipients.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
11. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a known history of Human Immunodeficiency Virus (HIV) infection.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
17. Has had an allogenic tissue/solid organ transplant.
18. Child-Pugh class B or C cirrhosis of liver.
19. Patients with a history of selective internal radiation therapy (eg, microsphere radioembolization) or who have received radiotherapy to the abdominal area prior to the initiation of study treatment.
20. Patients who have an inadequate hepatic reserve, as judged by the investigator; ie, normal liver tissue volume <700 mL.
21. Patients who fail to follow the radiation dose constraint of any critical organ.
22. Has a preexisting Grade ≥3 gastrointestinal or non-gastrointestinal fistula.
23. Has clinically significant hemoptysis from any source or tumor bleeding within 2 weeks prior to the first dose of study intervention.
24. Has significant cardiovascular impairment within 12 months prior to the first dose of study intervention such as history of congestive heart failure greater than NYHA Class II, unstable angina, myocardial infarction or cerebrovascular accident stroke, or cardiac arrhythmia associated with hemodynamic instability.
25. Has had major surgery to the liver within 4 weeks prior to the first dose of study intervention.

    Note: f participant underwent major surgery, they must have adequately recovered from the toxicity and/or complications from the intervention prior to starting study intervention.
26. Has had a minor surgery (ie, simple excision) within 7 days prior to the first dose of study intervention (Cycle 1 Day 1).
27. Has serious nonhealing wound, ulcer, or bone fracture.
28. Participants with proteinuria >1+ on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein ≥1 g/24 hours will be ineligible.
29. Has prolongation of corrected QT (QTc) interval to >480 ms (corrected by Fridericia Formula) or is taking drugs known to prolong the QT interval, including Class Ia and III antiarrhythmics (Quinidine, Procainamide, Disopyramide, Amiodarone, Sotalol, Ibutilide, Dofetilide & Dronedarone).
30. Has LVEF below the institutional normal range as determined by MUGA or echocardiogram (ECHO).
31. Has dual active HBV infection (HbsAg positive and /or detectable HBV DNA) and HCV infection (anti-HCV Ab positive and detectable HCV RNA) at study entry.
32. Uncontrolled blood pressure > 140/90 mmHg in spite of an optimal regimen of antihypertensive medication.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
safety rate | The period to evaluate DLT is for 28 days after completion of SBRT.
  In stage 0 and stage I interim analysis DLT will be assessed after 3 patients for each stage are accrued to the study. In stage II interim analysis for 6 (from stage 0 and I) + 6 (from stage II) patients, ≤4 patients with DLT and ≥6 patients with CR/PR are the criteria for stage III patient accrual.
objective response rate | From date of study intervention to 2.5 years
  Tumor measurements and response evaluations are conducted by an independent radiologist based on liver dynamic CT or MRI images at screening and every follow-up image after allocation. A second radiologist will perform an independent blinded image review at the end of the study without interfering with the primary judgment concerning disease progression and treatment decision. The response evaluation criteria are according to mRECIST.

SECONDARY OUTCOMES:
Progression-free survival and overall survival | From date of study intervention to 2.5 years
  Survival outcomes are calculated from date of allocation. Progression is defined as progressive disease by mRECIST or death from any cause. Overall survival is the time from allocation to death from any cause. Survival curves are determined by the Kaplan-Meier method.

OTHER OUTCOMES:
Immune biomarkers | From date of study intervention to 2.5 years
  1. Pre-treatment tumor tissue (i.e., biopsy or prior surgery) or blood sample is mandatory for biomarker study accompanying the clinical trial.
  2. The collected biomarkers will be analyzed for the correlation with the response of portal vein tumor thrombosis, progression-free survival, and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsien Cheng, Principal Investigator — Department of Internal Medicine, NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiawn, Taiwan

IPD SHARING:
Plan to Share IPD: No